CLINICAL TRIAL: NCT00526019
Title: Characteristics of Symptomatic Asthma Remissions
Brief Title: Persistence of Airway Inflammation and Remodeling in Subjects With Symptomatic or Complete Asthma Remission
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Louis-Philippe Boulet, MD, FRCPC, FCCP, Laval University
Other Study IDs: HL-07-20088
Record Dates: First submitted 2007-09-05; First posted 2007-09-06 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Asthma
Keywords: remission of asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Complete remission of their asthma: Subjects in complete remission of their asthma Subjects in complete remission of their asthma: absence of respiratory symptoms, no rescue asthma medication need and an optimal pulmonary function and normal PC20 methacholine (>16 mg/ml) for more than two years (with no current treatment).
- Symptomatic remission ofasthma: Subjects in symptomatic remission of their asthma (No asthma symptoms in the last 2 years, no asthma medication, PC20 methacholine <16 mg/ml)
- Current asthma (mild asthma): Subjects with current asthma (Mild asthma)
- Healthy controls: Healthy controls

SUMMARY:
This study aims at determining the patterns of asthma remission, the prevalence of these different patterns, the various factors associated with such remissions and possible recurrences of asthma, in order to determine the mechanisms involved in these processes.

The investigators therefore want to document these specificities in subjects in complete remission of their asthma, and those in only symptomatic remission of their asthma, in comparison with mildly symptomatic asthmatic subjects and healthy controls.

DETAILED DESCRIPTION:
Primary Outcome Measures :

* Airway inflammation (% induced sputum eosinophils)

Secondary Outcome Measures:

* Perception of induced respiratory symptoms
* Airway response to methacholine and AMP, and perception scores
* Diurnal variation in Peak Expiratory Flows
* Profile of regulatory T cells in the peripheral blood
* Changes in these parameters over time (baseline, 6 months, 1 and 2 years)

ELIGIBILITY:
Inclusion Criteria:

* In remission of their asthma: absence of respiratory symptoms, no rescue asthma medication need and (for complete remission) an optimal pulmonary function (FEV1 > 90%) and normal PC20 methacholine for more than two years (with no current treatment).
* With a proven past history of asthma from medical files (reversible airway obstruction (> 12% FEV1 after bronchodilator or 20% by other means) proven by spirometry, PEF measures or methacholine challenge according to current criteria + previous symptoms and asthma medication use), having no more asthma symptoms and not having used asthma medication for more than 2 years.
* Agree to sign the consent form.
* No other condition that could interfere with the study measurements.

Exclusion Criteria:

* Unable to adhere to the protocol requirements.
* Other current respiratory disease.
* Upper or lower respiratory tract infection or use of antibiotics < 1 month.
* Use of oral corticosteroids within the last 3 months.
* Signs or symptoms of progressive or uncontrolled renal, hepatic, hematologic, endocrine, pulmonary, cardiac, neurologic, or cerebral disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects wiil be offered to volunteer from advertisements in newspaper. Subjects with asthma or in remission of asthma from primary care clinics will be offered to participate.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2007-09; Primary Completion 2011-06 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Boulet, MD, Principal Investigator — Hôpital Laval